CLINICAL TRIAL: NCT04825587
Title: The Pediatric ALL Evaluation and Trial: A Randomized, Controlled Trial
Brief Title: The Pediatric ALL Evaluation and Trial
Acronym: PALLET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Texas Children's (Unknown); UCSF Benioff Children's Hospital - San Francisco (Unknown)
Responsible Party: Principal Investigator, Neeraj Patel, MD, MD, Orthopedic Surgery & Sports Medicine, Surgery, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-3610
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: ACL Injury; ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: The overall aim of this multicenter RCT is to determine whether concomitant ALL reconstruction in children undergoing and ACL reconstruction will result in a lower rate of graft failure than ACL reconstruction alone.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concomitant ACL and ALL reconstruction (Experimental): The participant will undergo both the ACL and ALL reconstruction surgery.
  Interventions: Procedure: Patients will be randomized into one of two study arms: (1) concomitant ACL and ALL reconstruction or (2) ACL reconstruction alone.
- ACL reconstruction alone (Experimental): The participant will undergo only ACL reconstruction surgery.
  Interventions: Procedure: Patients will be randomized into one of two study arms: (1) concomitant ACL and ALL reconstruction or (2) ACL reconstruction alone.

INTERVENTIONS:
Procedure: Patients will be randomized into one of two study arms: (1) concomitant ACL and ALL reconstruction or (2) ACL reconstruction alone. — By randomizing patients into one of two study arms: (1) concomitant ACL and ALL reconstruction or (2) ACL reconstruction alone, following statistical analysis, we hope to determine whether concomitant ALL reconstruction in children undergoing and ACL reconstruction will longitudinally result in a lower rate of graft failure than ACL reconstruction alone.

SUMMARY:
The overall aim of this multicenter RCT is to determine whether concomitant ALL reconstruction in children undergoing and ACL reconstruction will longitudinally result in a lower rate of graft failure than ACL reconstruction alone.

DETAILED DESCRIPTION:
Studies have reported a rising incidence of anterior cruciate ligament (ACL) injuries in children and adolescents. Beck et al reported a 2.3% annual increase between 1994 and 2013. In New York State, the rate of pediatric ACL reconstruction climbed from 17.6/100,000 in 1990 to 50.9/100,000 by 2009. Other reports echo these findings. After ACL reconstruction, children are known to be at a higher risk for complications than adults. For example, while the rate of postoperative graft failure in adults was 3% to 4% in large national registries, as many as 12% to 19% of pediatric patients may sustain graft rupture. This can have substantial medical, financial, and psychosocial implications on the patient and family. Additionally, the results of revision ACL reconstruction are, on average, worse than after index surgery. Exploration of treatments that may lower the rate of re-injury is paramount in this population that is at highest risk.

In the adult population, a growing number of studies have suggested that concomitant reconstruction of the anterolateral ligament (ALL) with the ACL may help lower this risk. The ALL was likely first characterized in 1879 by the French surgeon Segond, who commented on the presence of a "pearly, resistant, fibrous band" in the lateral aspect of the knee. However, only in 2012 was the structure given the name "anterolateral ligament" after it was consistently identified in cadaveric specimens. Some studies suggest that the ALL is damaged during anterior cruciate ligament (ACL) injury, implying that it may supplement the ACL in providing rotational and translational stability. Biomechanical studies have confirmed that it likely plays a role in rotational stability.

A number of ALL reconstruction techniques have been developed with the hope of lowering the rate of re-injury after ACL reconstruction. Early literature in the adult population suggests that this may indeed be the case. Early case series suggested that concomitant ALL reconstruction resulted in high rates of return to sport and a low ACL graft failure rate (2.6%). Comparative retrospective studies in adults suggest better patient reported outcome scores, meniscal repair healing, and rates of return to sports when the ALL is reconstructed with the ACL compared to isolated ACL reconstruction. Finally, a prospective cohort study of adults reported that hamstring autograft ACL reconstruction with concomitant ALL reconstruction resulted in 3.1 times lower odds of graft failure than isolated hamstring ACL reconstruction and 2.5 times lower odds of failure than isolated patellar tendon ACL reconstruction.

The hypotheses to be tested in this study have never been evaluated in the pediatric population. Furthermore, the proposed investigation is a randomized controlled trial, which will allow it to provide novel results with high-level evidence. The results of such a study have the potential to change practice in a meaningful, tangible way and affect the outcomes of thousands of children annually. In addition to the medical and functional impact, there could also be important financial and psychosocial implications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and under
* Surgery within 6 months of injury
* Undergoing primary ACL reconstruction without previous injury or surgery
* Quadriceps tendon autograft ACL reconstruction
* Closing or closed physes

Exclusion Criteria:

* Over 18 years old
* Previous ipsilateral knee injury or surgery
* Neuromuscular or developmental disorders affecting knee anatomy, cognition, or neuromuscular control
* Other concomitant ligament reconstruction aside from the ALL (i.e., MCL, PCL, PLC)
* Revision ACL reconstruction
* ACL reconstruction with graft other than quadriceps tendon
* IT band (modified MacIntosh) ACL reconstruction
* A cartilage lesion requiring anything more than debridement
* Open physes requiring both femoral and tibial physeal-sparing technique

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Graft failure | Complete when all 780 participants have been recruited, received an intervention and have been followed for data collection for up to 5 years.
  To determine whether concomitant ALL reconstruction in children undergoing and ACL reconstruction will longitudinally result in a lower rate of graft failure (confirmed graft re-tear or asymmetric, increased pivot shift) than ACL reconstruction alone.

SECONDARY OUTCOMES:
Complications of ALL reconstruction | Complete when all 780 participants have been recruited, received an intervention and have been followed for data collection for up to 5 years.
  To determine the rate and severity of complications related specifically to ALL reconstruction in children.
Patient reported outcome measures | Complete when all 780 participants have been recruited, received an intervention and have been followed for data collection for up to 5 years.
  To collect and compare patient reported outcome (PRO) scores (as measured by the Pedi-IKDC, Lysholm, HSS Pedi-FABS, and PROMIS surveys) in children undergoing ACL reconstruction alone, and children undergoing combined ACL and ALL reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Patel, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Lurie Children's Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Collected Participant info that may be collected and shared :Personal and health information, Past/present medical records, Records from study visits/phone calls. Behavioral or mental health info about the participants will be collected and may be shared.The study staff, employees, and Medical Staff of Lurie Children's may use participant's info for this study and share it with study sponsor, POSNA and those working with the sponsor, IRB, Participant's other providers and their staff directly involved in their care, if their provider is a part of the Lurie Children's electronic health information exchange: The Office of Human Research Protections (OHRP), the Food and Drug Administration (FDA), or other government offices. We cannot guarantee that those listed above will not share it with others without participant's permission. Participant's names will not be included in any written or verbal reports of study results.
Supporting Information: Study Protocol, ICF
Time Frame: from the study start up/participant recruitment (beginning April 2021) until 1/1/2030
Access Criteria: Study personnel only